CLINICAL TRIAL: NCT02366273
Title: Diabetes and Psoriasis: Study on Prevalence, Role of Inflammation and Insulin-resistance
Brief Title: Diabetes and Psoriasis
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, University of Pavia
Other Study IDs: P-20140023881
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; Psoriasis
Keywords: Diabetes; Psoriasis; Inflammation; Insulin-resistance
MeSH Terms: conditions — Diabetes Mellitus; Psoriasis; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PASI and HOMA index

SUMMARY:
Patients with psoriasis will be evaluated. The investigators will collect personal history, concomitant diseases and in particular the presence of type 2 diabetes mellitus, impaired fasting glucose and impaired glucose tollerance. The aim of the study will be to evaluate if there is a correlation among inflammation, insulin-resistance and psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* patients with psoriasis

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with psoriasis
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of correlation between diabetes and psoriasis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, FESC, Principal Investigator — University of Pavia - IRCCS Policlinico San Matteo Foundation
Locations (1):
- IRCCS Policlinico San Matteo Foundation, Pavia, Italy